CLINICAL TRIAL: NCT03629236
Title: A Multicenter, Prospective, Randomized, Open-Label Study With a Crossover Extension Option to Evaluate the Safety and Efficacy of GrafixPL for the Treatment of Chronic Venous Leg Ulcers
Brief Title: Study to Evaluate Safety and Efficacy of GrafixPL for the Treatment of Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osiris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Osiris Protocol 360; NCT03543007 (obsolete NCT alias)
Record Dates: First submitted 2018-05-18; First posted 2018-08-14 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-03

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GrafixPL (Experimental)
  Interventions: Other: GrafixPL
- Control (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: GrafixPL — Debridement, GrafixPL application, dressing application, standard compression therapy
  Other Names: Tissue Allograft
  Arms: GrafixPL
Other: Control — Debridement, dressing application, standard compression therapy
  Arms: Control

SUMMARY:
A Multicenter, Prospective, Randomized, Open-Label Study with a Crossover Extension Option to Evaluate the Safety and Efficacy of GrafixPL for the Treatment of Chronic VLUs

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older, as of the date of screening
2. An Index Ulcer that is chronic (defined as present for > 4 weeks, but not present for more than 52 weeks at Screening Visit 1)
3. Index Ulcer is located on the leg, below the knee and above the malleoli (ulcer may be inclusive of the malleoli)
4. The Index Ulcer is between 1 cm2 and 25 cm2, inclusive, at the Screening and Baseline Visits. The longest dimension of the index ulcer cannot exceed 10 cm at the Baseline Visit.
5. The Index Ulcer has had compression therapy for > 2 weeks at Screening Visit 1
6. The Index Ulcer extends into the dermis or subcutaneous tissue without evidence of exposed muscle, tendon, bone, or joint capsule
7. Patient has adequate circulation to the foot, as documented up to 14 days prior to Screening Visit 1
8. Confirmed diagnosis of venous insufficiency, as documented up to 30 days prior to enrollment

Exclusion Criteria:

1. Index Ulcer is of non-venous pathophysiology
2. Gangrene is present on any part of the affected limb
3. Patient is unable to tolerate standard compression therapy
4. Glycated hemoglobin A1c (HbA1c) level of > 14% in any patient with type 1 or type 2 diabetes mellitus, as documented up to 14 days prior to Screening Visit 1
5. Patient is receiving intravenous (IV) corticosteroids, immunosuppressive or cytotoxic agents at any time during the screening period
6. Patient has an ulcer within 5 cm of the Index Ulcer identified for study consideration
7. Patient is Human Immunodeficiency Virus (HIV) positive or has Acquired Immune Deficiency Syndrome (AIDS)
8. Current evidence of infection at the Index Ulcer, including cellulitis and/or pus drainage from the ulcer site at the time of Screening and Baseline Visits
9. Evidence of osteomyelitis at the time of Screening and Baseline Visits
10. Patient has active malignancy other than non-melanoma skin cancer
11. Patient's Index Ulcer has decreased by ≥ 30% between Screening Visit 1 and the Baseline Visit during the screening period
12. Patient has untreated alcohol or substance abuse at the time of Screening Visit 1
13. Pregnant women and women who are breastfeeding
14. Patient is currently enrolled in or has participated in another investigational device, drug, or biological trial within 30 days prior to Screening Visit 1
15. Patient has had within 14 days of Screening Visit 1, or is currently undergoing, or is planning for ulcer treatments with growth factors, living skin, dermal substitutes or other advanced biological therapies
16. Patient is an employee, or an immediate family member of an employee, of the sponsor company or site research staff conducting the study
17. Patients who have already been randomized in Protocol 360 at any center may not be considered for screening or for re-entry into the trial at any center, even after the End of Treatment Study Visit
18. Patients with a history of poor compliance, or an unwillingness or inability to adhere to the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Complete closure of the index ulcer | Up to 84 days after the Baseline Visit

SECONDARY OUTCOMES:
Time to initial ulcer closure | Up to 84 days after the Baseline Visit
Measurement of percent area reduction in ulcers that do not achieve closure | 84 days after the Baseline Visit
Proportion of patients with ulcer reoccurrence in Follow-Up Phase | Up to 6 months after initial ulcer closure
Proportion of patients in the Crossover Extension Treatment Phase who achieve complete ulcer closure | Up to 91 days after initial Treatment Phase
Time to initial ulcer among patients in the Crossover Extension Treatment Phase | Up to 91 days after initial Treatment Phase

OTHER OUTCOMES:
Number and type of AEs and SAEs | Through study completion, approximately 38 weeks
Number and type of ulcer related complications | Through study completion, approximately 38 weeks
CWIS Questionnaire | Through study completion, approximately 38 weeks
WPAI Questionnaire | Through study completion, approximately 38 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Banerjee, PHD, Study Chair — Smith & Nephew, Inc.
Locations (2):
- United States (2):
  - Integral Clinical Trial Solutions, Doral, Florida
  - SSH, Weymouth, Massachusetts

REFERENCES:
- [Derived] Dhillon Y, Levine L, Tovmassian G, Reyzelman A, Perez-Clavijo F, Wodie F, Cazzell S, Grossman A, Robinson L, Sigal F, Kirsner RS, Vartivarian M, Saunders M, Banerjee J. A Multicenter, Randomized, Controlled, Clinical Trial Evaluating a Lyopreserved Amniotic Membrane in the Treatment of Venous Leg Ulcers. Health Sci Rep. 2025 May 4;8(5):e70819. doi: 10.1002/hsr2.70819. eCollection 2025 May. PMID 40330756